CLINICAL TRIAL: NCT04769635
Title: Impact of Continuous Positive Airway Pressure Therapy on Pulmonary Hypertension and Exercise Capacity in Newly Diagnosed Obstructive Sleep Apnea Patients
Brief Title: CPAP Therapy in Obstructive Sleep Apnea Patients With Pulmonary Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Ahmad Abbas, Lecturer of chest diseases, Zagazig University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZU-IRB#5654
Record Dates: First submitted 2021-02-20; First posted 2021-02-24 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- CPAP ttt (Experimental)
  Interventions: Device: CPAP therapy

INTERVENTIONS:
Device: CPAP therapy — All studied patients were received CPAP therapy with average cumulative adherence ⩾4 h/day of >70% nights [380] obtained from device download with AHI<5 /hr

SUMMARY:
All patients are newly diagnosed Obstructive Sleep Apnea patients performing full night polysmnographic sleep study, whose echocardiographic findings elucidate presence of pulmonary hypertension(PH). These patients seemed to have PH if mPAP ≥25 mmHg . All studied patients were received CPAP therapy with average cumulative adherence ⩾4 h/day of >70% nights [380] obtained from device download with AHI<5 /hr

Echocardiography:

It was performed initially to diagnose pulmonary hypertension and repeated after three months of CPAP therapy as a follow up . All enrolled patients were subjected to trans-thoracic echocardiography using Ultrasound system (Vivid I, GE Healthcare, Little Chalfont, UK), with a 2.5 MHz transducer. Certain measurements were then used to calculate mPAP.

Patients were considered to have PH if mPAP ≥25 mmHg, and were classified into mild (20-40 mmHg), moderate (41-55 mmHg), and severe (>55 mmHg) degrees.

Evidence of PH is found by Doppler echocardiography showing an elevated right ventricular systolic pressure (RVSP).

ELIGIBILITY:
Inclusion Criteria:

All patients are newly diagnosed Obstructive Sleep Apnea patients performing full night polysmnographic sleep study, whose echocardiographic findings elucidate presence of pulmonary hypertension(PH).

Exclusion Criteria:

* Patients aged < 18 years
* Patients with secondary PH, due to pulmonary diseases, or left ventricular heart diseases , or chronic thromboembolic disorders.
* Patients on long term oxygen therapy (LTOT).
* Patients with respiratory neuromuscular weaknesses or chest wall deformities.
* End-organ failure and malignancies
* Obesity hypoventilation syndrome.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2020-04-20 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
change of mean pulmonary artery pressure measured by echo | 3 months

SECONDARY OUTCOMES:
Exercise capacity improvement measured by six minute walking test | 3 months
Exercise capacity improvement measured by maximun o2 consumption | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmad Abbas, Zagazig, Sharqia Province, Egypt